CLINICAL TRIAL: NCT05986149
Title: Making Intergenerational Connections Through Arts
Status: Recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Hon K. Yuen, PhD, Professor, University of Alabama at Birmingham
Other Study IDs: IRB-300008546
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Older Adults
MeSH Terms: interventions — Culture Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Conversation about arts and culture — intergenerational conversation about arts and culture between older adults and international students who native language is not English.

SUMMARY:
The purpose of the study is to evaluate the impact on older adults' wellbeing of participating in a 10-week conversation about arts and culture with an international university student whose native language is not English.

DETAILED DESCRIPTION:
Older adults residing in subsidized housing will participate in a series of online conversations over 10 weeks about various arts and culture with an international university student enrolled at the University of Alabama at Birmingham (UAB); each weekly session will last for about 30 min to one hour.

Participants will complete survey questionnaires before and after the 10-week conversation program, and an exit interview at the end of the conversation program.

ELIGIBILITY:
Inclusion Criteria:

1. Live alone
2. older than 60 years old
3. Residence in a subsidized apartment for at least one year
4. Able to carry on a daily conversation with or without hearing aids
5. Intact cognition as indicated by a score of greater than 5 on the Short Portable Mental Status Questionnaire (SPMSQ)
6. have a working smart phone that can do video-conferencing
7. being able to provide informed consent

Exclusion Criteria:

1. having physical, or sensory (visual or hearing) deficits or language barriers (non-English communicators) that may impede study participation
2. non-English speaker

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: residents living in low income housing
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
University of California, Los Angeles (UCLA) Loneliness Scale | baseline
  (ULS-8, Hays & Dimatteo, 1987) measures one's subjective feelings of loneliness as well as feelings of social isolation. It has 8 items rated on a 4-level frequency score scale (0=never to 3=always) with higher scores indicating a higher degree of loneliness. Some items require reverse scoring.
University of California, Los Angeles (UCLA) Loneliness Scale | at 10 weeks
  (ULS-8, Hays & Dimatteo, 1987) measures one's subjective feelings of loneliness as well as feelings of social isolation. It has 8 items rated on a 4-level frequency score scale (0=never to 3=always) with higher scores indicating a higher degree of loneliness. Some items require reverse scoring.
University of California, Los Angeles (UCLA) Loneliness Scale | at 2 months
  (ULS-8, Hays & Dimatteo, 1987) measures one's subjective feelings of loneliness as well as feelings of social isolation. It has 8 items rated on a 4-level frequency score scale (0=never to 3=always) with higher scores indicating a higher degree of loneliness. Some items require reverse scoring.
De Jong Gierveld Loneliness Scale | baseline
  De Jong Gierveld Loneliness Scale - 6 items) measures one's emotional loneliness (lack of intimate relationship, 3 items) and social loneliness (lack of wider social network, 3 items). There are negatively (1-3) and positively (4-6) worded items. On the negatively worded items, the neutral and positive answers are scored as "1". Therefore, on questions 1-3 score Yes=1, More or less=1, and No=0. On the positively worded items, the neutral and negative answers are scored as "1". Therefore, on questions 4-6, score Yes=0, More or less=1, and No=1. This gives a possible range of scores from 0 to 6, with 0=least lonely, and 6=most lonely.
De Jong Gierveld Loneliness Scale | at 10 weeks
  De Jong Gierveld Loneliness Scale - 6 items) measures one's emotional loneliness (lack of intimate relationship, 3 items) and social loneliness (lack of wider social network, 3 items). There are negatively (1-3) and positively (4-6) worded items. On the negatively worded items, the neutral and positive answers are scored as "1". Therefore, on questions 1-3 score Yes=1, More or less=1, and No=0. On the positively worded items, the neutral and negative answers are scored as "1". Therefore, on questions 4-6, score Yes=0, More or less=1, and No=1. This gives a possible range of scores from 0 to 6, with 0=least lonely, and 6=most lonely.
De Jong Gierveld Loneliness Scale | at 2 months
  De Jong Gierveld Loneliness Scale - 6 items) measures one's emotional loneliness (lack of intimate relationship, 3 items) and social loneliness (lack of wider social network, 3 items). There are negatively (1-3) and positively (4-6) worded items. On the negatively worded items, the neutral and positive answers are scored as "1". Therefore, on questions 1-3 score Yes=1, More or less=1, and No=0. On the positively worded items, the neutral and negative answers are scored as "1". Therefore, on questions 4-6, score Yes=0, More or less=1, and No=1. This gives a possible range of scores from 0 to 6, with 0=least lonely, and 6=most lonely.
Social Connectedness Scale (SCS) | baseline
  It has 8 items rated on a 6-point Likert-type scale (1=strongly agree to 6=strongly disagree) with higher scores indicating a more reported sense of social connectedness and belongingness.
Social Connectedness Scale (SCS) | at 10 weeks
  It has 8 items rated on a 6-point Likert-type scale (1=strongly agree to 6=strongly disagree) with higher scores indicating a more reported sense of social connectedness and belongingness.
Social Connectedness Scale (SCS) | at 2 months
  It has 8 items rated on a 6-point Likert-type scale (1=strongly agree to 6=strongly disagree) with higher scores indicating a more reported sense of social connectedness and belongingness.
Medical Outcomes Study Social Support Survey (MOSSS) | baseline
  It has 3 items rated on a 5-point Likert-type scale ( 'none of the time' = 1 to 'all of the time' = 5) with higher scores indicating a more positive social interaction.
Medical Outcomes Study Social Support Survey (MOSSS) | at 10 weeks
  It has 3 items rated on a 5-point Likert-type scale ( 'none of the time' = 1 to 'all of the time' = 5) with higher scores indicating a more positive social interaction.
Medical Outcomes Study Social Support Survey (MOSSS) | at 2 months
  It has 3 items rated on a 5-point Likert-type scale ( 'none of the time' = 1 to 'all of the time' = 5) with higher scores indicating a more positive social interaction.

SECONDARY OUTCOMES:
Satisfaction with Life Scale (SWLS) | baseline
  SWLS (Diener et al., 1985) is used to evaluate the global self-assessment of one's quality of life. The SWLS consists of five statements where participants indicated how much they agreed or disagreed with each statement about their life satisfaction using a 7-point Likert scale, ranging from 1 = strongly disagree to 7 = strongly agree. Higher scores indicate more satisfaction with one's life.
Satisfaction with Life Scale (SWLS) | at 10 weeks
  SWLS (Diener et al., 1985) is used to evaluate the global self-assessment of one's quality of life. The SWLS consists of five statements where participants indicated how much they agreed or disagreed with each statement about their life satisfaction using a 7-point Likert scale, ranging from 1 = strongly disagree to 7 = strongly agree. Higher scores indicate more satisfaction with one's life.
Satisfaction with Life Scale (SWLS) | at 2 months
  SWLS (Diener et al., 1985) is used to evaluate the global self-assessment of one's quality of life. The SWLS consists of five statements where participants indicated how much they agreed or disagreed with each statement about their life satisfaction using a 7-point Likert scale, ranging from 1 = strongly disagree to 7 = strongly agree. Higher scores indicate more satisfaction with one's life.
Warwick-Edinburgh Mental Well-being Scale (WEMWBS) | baseline
  The WEMWBS is intended to measure a person's functioning aspects of mental well-being (Stranges et al., 2014). The scale consists of 14 items, with each item rated on a 5-point Likert-type scale (1 = none of the time to 5 = all of the time). The total scores range from 14 to 70, with higher scores indicating greater mental well-being.
Warwick-Edinburgh Mental Well-being Scale (WEMWBS) | at 10 weeks
  The WEMWBS is intended to measure a person's functioning aspects of mental well-being (Stranges et al., 2014). The scale consists of 14 items, with each item rated on a 5-point Likert-type scale (1 = none of the time to 5 = all of the time). The total scores range from 14 to 70, with higher scores indicating greater mental well-being.
Warwick-Edinburgh Mental Well-being Scale (WEMWBS) | at 2 months
  The WEMWBS is intended to measure a person's functioning aspects of mental well-being (Stranges et al., 2014). The scale consists of 14 items, with each item rated on a 5-point Likert-type scale (1 = none of the time to 5 = all of the time). The total scores range from 14 to 70, with higher scores indicating greater mental well-being.
Patient Health Questionnaire - 9 items (PHQ-9) | baseline
  is to measure for depression, where participants are asked to rate how often they were bothered by specific symptoms over the last two weeks. It has 9 items rated on a 4-level frequency score scale (0=not at all to 3=nearly every day) with higher scores indicating greater symptoms of depression.
Patient Health Questionnaire - 9 items (PHQ-9) | at 10 weeks
  is to measure for depression, where participants are asked to rate how often they were bothered by specific symptoms over the last two weeks. It has 9 items rated on a 4-level frequency score scale (0=not at all to 3=nearly every day) with higher scores indicating greater symptoms of depression.
Patient Health Questionnaire - 9 items (PHQ-9) | at 2 months
  is to measure for depression, where participants are asked to rate how often they were bothered by specific symptoms over the last two weeks. It has 9 items rated on a 4-level frequency score scale (0=not at all to 3=nearly every day) with higher scores indicating greater symptoms of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Hon K Yuen, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No